CLINICAL TRIAL: NCT04709341
Title: Optimization of Transradial-Band Removal Following Transradial Arterial Access for Interventional Radiology Diagnostic and Interventional Procedures (A Pilot Study)
Brief Title: Transradial-Band Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00088481
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Radial Artery Incision Site Closure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Experimental)
  Interventions: Device: TR Band 60MIN
- Group B (Active Comparator)
  Interventions: Device: TR Band 120MIN

INTERVENTIONS:
Device: TR Band 60MIN — TR-Band will be in left in place for 15 minutes before it is gradually deflated by 25% at 15 minute intervals
  Arms: Group A
Device: TR Band 120MIN — TR-Band is left in place for 60 minutes before it is gradually deflated by 25% at 15 minute intervals
  Arms: Group B

SUMMARY:
In the study group, the TR-Band will be in left in place for 15 minutes before it is gradually deflated by 25% at 15 minute intervals. In the standard of care group, the TR-Band is left in place for 60 minutes before it is gradually deflated by 25% at 15 minute intervals. The aim of the study is to reduce the time the device is in place while minimizing potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Have an acceptable Barbeau test (i.e. type A through C)
* Have acceptable coagulation parameters (based on PT, INR, platelet count, and appropriate pre-procedural management of anticoagulants, See Table 1)
* The caliber of the left radial artery based on a pre-procedure sonographic evaluation will need to be greater than or equal to 1.6 mm.
* The appropriate pre-procedural management of anticoagulants is based on the consensus guidelines established by Patel et al16.
* INR less than 1.5
* Platelet count greater than 50,000 platelet/uL
* Prothrombin time less than 15 seconds

Exclusion Criteria:

* If there is an unacceptable risk of bleeding diathesis, or
* If he or she is not a suitable candidate for transradial access based on a Barbeau test type D or a diameter of the left radial artery less than 1.6 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at MUSC's VIR Department, including University Hospital and outpatient clinics. Patients scheduled for angiographic procedures were screened for eligibility via Barbeau tests, ultrasounds, and lab reviews. Informed consent was obtained during consultations or in recovery bays. Recruitment involved 30 randomized patients divided into expedited and standard protocol groups.
Pre-assignment Details: No significant events, such as washout or run-in periods, occurred after participant enrollment and before group assignment. All participants who met eligibility criteria, including acceptable Barbeau test results, ultrasound evaluation, and coagulation parameters, were randomized directly into the expedited or standard protocol groups. No exclusions were reported after enrollment and prior to randomization
Period: Overall Study
Arm/Group | Group A | Group B
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included 30 patients randomized into expedited (n=15) and standard (n=15) protocol groups. All participants met inclusion criteria: age >18 years, Barbeau test types A-C, radial artery diameter ≥1.6 mm, and acceptable coagulation parameters (platelet count >50,000/µL, INR <1.5, PT <15s). No significant differences in demographics or clinical characteristics were observed between groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (16.67) | 64.2 (11.7) | 62.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Bleeding
Description: Continued ooze requiring re-inflation of the TR-Band or subcutaneous ecchymosis without a discernable hematoma
Time Frame: an average of 12 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 15 | 15
Participants | 0 | 1

2. Primary Outcome: Percentage of Participants With Bleeding
Description: Continued ooze requiring re-inflation of the TR-Band or subcutaneous ecchymosis without a discernable hematoma
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 15 | 15
Participants | 0 | 1

3. Primary Outcome: Left Radial Artery Occlusion
Description: Reduced or absence of radial artery blood flow based on ultrasound and Barbeau test
Time Frame: 30 days post procedure
Population: No patients presented with this symptom during the TR Band Procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: The outcomes focus on safety, efficacy, and complications specific to the radial artery access site, and no deaths were mentioned or attributed to the procedures or protocols
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=15) | Group B (N=15)
Mild Bruising (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT04709341/Prot_SAP_000.pdf